CLINICAL TRIAL: NCT00585858
Title: Cytokine Kinetics Assay to Assess the Presence or Absence of Tolerance in Organ Transplant Recipients
Brief Title: Cytokine Kinetics Test to Assess the Presence or Absence of Tolerance in Organ Transplant
Status: Terminated | Type: Observational
Why Stopped: PI leaving institution
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: H-2006-0437
Record Dates: First submitted 2007-12-26; First posted 2008-01-03 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Kidney Transplantation; Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Subjects on mimimal or no immunosuppression and no rejection history
- 2: Subjects who have had rejection on conventional immunosuppression
- 3: Subjects who have not had acute or chronic rejection who are on conventional immunosuppression

SUMMARY:
The purpose of this pilot study is to determine if there is clinical correlation between the CKT and transplant recipients who are known to be on minimal or no immunosuppression (presumed tolerant) and those who are on conventional amounts of immunosuppression and have either experienced rejection (presumed hyper-responsive to donor) or have not experienced rejection (unknown responsive state).

ELIGIBILITY:
Inclusion Criteria:

* Kidney or liver transplant recipients for whom donor cells are available

Exclusion Criteria:

* HcT <32%

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Kidney or liver transplant recipients
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2006-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Correlation between cytokine kinetics test and clinical status of subject | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No